CLINICAL TRIAL: NCT06413940
Title: Effect of Mobile-health and Comprehensive Physical Therapy on Moderate-to-severe Obstructive Sleep Apnea Hypoventilation Syndrome
Brief Title: Exploring the Clinical Efficacy of Remote Management Applications Through Comprehensive Physical Therapy for Patients With Moderate to Severe Sleep Apnea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-ZX036
Record Dates: First submitted 2024-04-26; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: OSAHS; Oropharyngeal Muscle Training; Aerobic Exercise; Comprehensive Physical Therapy; M-health
Keywords: OSAHS; Comprehensive physical therapy; m-health
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Myofunctional Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Subjects in the control group will receive usual care(On-site healthy lifestyle promotion)
- Physical therapy group (Experimental): Subjects in the physical therapy group will receive myofunctional therapy and inspiratory muscle training
  Interventions: Behavioral: Myofunctional Therapy; Behavioral: Inspiratory Muscle Training
- Combined Exercise Group (Experimental): Subjects in the combined exercise group will receive myofunctional therapy ,inspiratory muscle training and aerobic training
  Interventions: Behavioral: Myofunctional Therapy; Behavioral: Inspiratory Muscle Training; Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Myofunctional Therapy — Oropharyngeal and tongue exercises : strengthening upper airway muscle 20 minutes
  Other Names: MT
  Arms: Combined Exercise Group; Physical therapy group
Behavioral: Inspiratory Muscle Training — Respiratory muscle strengthening:inspiratory muscle strengthening by resistive loading of 50% maximum inspiratory pressure.
  Other Names: IMT
  Arms: Combined Exercise Group; Physical therapy group
Behavioral: Aerobic Exercise — Exercise intensity :40%-60% HRmax , 3-5 days/week
  Other Names: AE
  Arms: Combined Exercise Group

SUMMARY:
To observe comprehensive physical therapy program for OSAHS patients

DETAILED DESCRIPTION:
This study proposes to conduct a randomized controlled trial ，using an APP and wearable devices to provide comprehensive physical therapy and monitoring for people with moderate to severe OSAHS,to assess the effectiveness and adherence of different physiotherapy programs for patients with moderate-to-severe OSAHS by observing the improvement of sleep apnea hypoventilation index (AHI), nocturnal minimum oxygen saturation (Low SpO2), mean oxygen saturation (Mean SpO2), and other health outcomes in the study population. It is expected to explore a clinical treatment pathway suitable for patients with moderate-to-severe OSAHS through mobile app and comprehensive physical therapy, improve the treatment adherence of OSAHS patients, enhance the level of health management services in hospitals, and obtain more physical health and health economic benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 60 years;
2. Those who have been recently diagnosed with moderate-to- severe OSAHS (AHI ≥ 15 beats/h) and who refuse or cannot tolerate the counter-adverse effects and refuse CPAP therapy after conventional medical advice;
3. Those who have not undergone any physical therapy;
4. Have some communication and comprehension skills and can use a smart phone;
5. Signed informed consent.

Exclusion Criteria:

1. BMI > 35kg/m2;
2. Patients with central and mixed sleep apnea;
3. Those who use sleep aids (including benzodiazepines and non-benzodiazepine sedative-hypnotics, anxiolytics with sleep-aiding effects, antidepressants, antipsychotics) and/or nutritional supplements;
4. Those suffering from acute myocardial infarction, acute tachyarrhythmia, pulmonary edema, severe aortic stenosis and other acute cardiovascular diseases;
5. Those with severe respiratory diseases such as asthma, chronic obstructive pulmonary disease (COPD), lung volume limitation (due to obesity, pregnancy, or spinal deformity), or cystic fibrosis, pneumothorax, or alveoli;
6. Those with hypothyroidism;
7. Those with severe ENT disorders such as severe upper airway obstruction (complete nasal congestion, tonsil grade III/IV), tongue-tie (Marchesani's protocol), motor symptoms limiting the tongue, antecedent or presence of temporomandibular joint disorders, and severe craniofacial injuries;
8. Those with inflammation-related systemic diseases (e.g., arthritis, tuberculosis, vasculitis, lupus);
9. Those who suffer from neuromuscular diseases (e.g., Duchenne muscular dystrophy) or diseases of the skeleton that prevent them from performing parallel movements due to exercise;
10. Those who smoke and drink alcohol;
11. Those who have had other sleep apnea treatments within 6 months (e.g., surgical procedures, MAD or CPAP treatments) that may affect the study results;
12. Ongoing clinical trials of drugs or devices in which they are participating;
13. Refusal to sign the informed consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
apnea-hypopnea index(AHI) | 3 months
  The home sleep apnea test (HSAT) device was used to detect the AHI of OSAHS patients, and the AHI was defined as the average number of apneas or hypoventilation per hour during sleep. According to the guidelines and related literature grouping,AHI ≥ 5 times/h was diagnosed as OSAHS, 5 times/h ≤ AHI < 15 times/h as mild OSAHS, and AHI ≥ 15 times/h as moderate to severe OSAHS.
  Our study observe the changes in apnea-hypopnea index from baseline to 3 months

SECONDARY OUTCOMES:
Minimum oxygen saturation at night（Low SpO2） | 3 months
  The home sleep apnea test (HSAT) device was used to detect the Low SpO2 of OSAHS patients. Our study observe the changes in Low SpO2 from baseline to 3 months.

OTHER OUTCOMES:
Peak oxygen uptake | 3 months
  Our study observe the changes in cardiorespiratory function from baseline to 3 months.In this program, a cycling graded incremental exercise program (Ramp program) was used, peak oxygen uptake was monitored.
Sleep quality | 3 months
  Changes in sleep quality from baseline to 3 months. The sleep quality was assessed by the Pittsburgh Sleep Quality Index (PSQI) .The scoring criteria are: 0-5 for very good sleep quality, 6-10 for okay sleep quality, 11-15 for average sleep quality, and 16-21 for very poor sleep quality, with higher total scores indicating poorer sleep quality;
Body composition | 3 months
  Changes in body composition analysis from baseline to 3 months.Using bioelectrical impedance analysis to monitor body weight,weight and height will be combined to report BMI in kg/m^2.
Quality of life score | 3 months
  Changes in quality of life from baseline to 3 months.Quality of life was assessed using the short form 36 questionnaire (SF-36).The score is 0-100, with higher scores indicating higher quality of patient survival.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Feng, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital